CLINICAL TRIAL: NCT00361816
Title: Human MATER and Idiopathic Infertility
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020195; 02-CH-0195
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-29

CONDITIONS: Infertility
Keywords: Maternal Effect Gene; Embryonic Development; Infertility
MeSH Terms: conditions — Infertility

SUMMARY:
Approximately 15 percent of couples experience infertility, yet no abnormalities can be detected in the man or the woman. In a number of couples, their embryos unexpectedly slow down growth or stop growth completely. Some of these situations may be genetically determined. For instance, a portion of cases may be caused by poor egg quality related to genetic or functional deficiencies in heretofore unidentified human maternal effect genes. A model has been developed of such unexplained fertility by creating a mouse line lacking a critical maternal effect gene. (Maternal effect genes produce mRNA or proteins that accumulate in the egg and are required for normal early embryonic development.) This pilot project will test the hypothesis that a similar defect may be a cause of human infertility.

Thirty cubic centimeters of blood will be collected from 40 women who have a clinical history consistent with a defective maternal effect gene. DNA from these blood cells will be examined and stored. Some of the blood cells will be treated so that they can be frozen and grown in the laboratory to produce more DNA in the future. If certain mutations are not found, that means that the prevalence of such mutations is less than 10 percent, and investigators may initiate another study with 100 women. If a common mutation is found in at least four patients, the investigators will seek to collect DNA from 150 normal fertile control women for comparison.

This project is purely investigational; therefore, findings will not be shared with participants.

...

DETAILED DESCRIPTION:
The pilot investigation will examine the hypothesis that human infertility may be caused by mutations in the human MATER gene. We will determine the prevalence of these mutations in a select group of women who have a clinical infertility history consistent with a possible defect in a maternal effect gene. After obtaining informed consent and DNA from 100 women, relevant mutations in the MATER gene will be searched for by single strand conformation polymorphism analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women to be included in this study will have a clinical infertility history that would be consistent with a possible defect in a maternal effect gene.

This includes women who meet the following criteria:

1. a clinical diagnosis of infertility,
2. never been pregnant, and
3. undergone treatment by in vitro fertilization and had at least 8 fertilized eggs as part of at least one in vitro fertilization cycle that failed to lead to a clinical pregnancy.

Women who have subsequently achieved a pregnancy by egg donation will be included.

Women of any age are eligible as long as they have otherwise met the inclusion criteria.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-05-03; Study Completion 2011-03-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Collins JA, Crosignani PG. Unexplained infertility: a review of diagnosis, prognosis, treatment efficacy and management. Int J Gynaecol Obstet. 1992 Dec;39(4):267-75. doi: 10.1016/0020-7292(92)90257-j. PMID 1361459
- [Background] Greenhouse S, Rankin T, Dean J. Genetic causes of female infertility: targeted mutagenesis in mice. Am J Hum Genet. 1998 Jun;62(6):1282-7. doi: 10.1086/301893. No abstract available. PMID 9585621
- [Background] Schultz RM. Regulation of zygotic gene activation in the mouse. Bioessays. 1993 Aug;15(8):531-8. doi: 10.1002/bies.950150806. PMID 8135766